CLINICAL TRIAL: NCT01290562
Title: A University of Toronto Phase II Study to Determine Efficacy of Stereotactic Body Radiotherapy (SBRT) for Spinal/Para-Spinal Metastases
Brief Title: Stereotactic Body Radiotherapy (SBRT) for Spinal/Para-Spinal Metastases (Spine SBRT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB 10-0540-C
Record Dates: First submitted 2011-02-03; First posted 2011-02-07 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Spinal Metastases
Keywords: SBRT; spinal Metastases; Paraspinal Metastases; spinal Metastases and SBRT; Paraspinal Metastases and SBRT
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stereotactic Body Radiotherapy (SBRT) (Experimental): Cohort 1: Patients with spinal metastases and no prior radiation Cohort 2: Patients with spinal metastases in a previously radiated field Cohort 3: Post-operative patients with spinal metastases
  Interventions: Radiation: Stereotactic Body Radiotherapy (SBRT)

INTERVENTIONS:
Radiation: Stereotactic Body Radiotherapy (SBRT) — One or more high dose(s) of radiation to treat the tumour.

SUMMARY:
Patients with new or recurrent spine metastases are currently treated with low doses of radiation delivered in up to ten treatments (wide-field radiation therapy). Stererotactic body radiotherapy (SBRT) is a technique in which high doses of radiation targeted precisely to the metastases to be treated are administered in a small number of sessions, thus reducing the radiation damage to the surrounding tissue and areas of the spine.

The purpose of this study is to evaluate the efficacy of spine SBRT as an alternative to conventional radiation for patients with no prior radiation, prior radiation, and in the post-operative patient

DETAILED DESCRIPTION:
Spine SBRT is currently being practiced as an alternative to conventional wide-field radiation in the up-front management of spinal metastases, in the re-irradiation scenario, and in the post-operative setting. This study proposes to treat patients with a uniform spine SBRT approach, and collect prospective outcome data as a basis for future randomized trial design. Preliminary evaluation of our technique has yielded acceptable accuracy in treatment delivery as compared to the literature, and our practice follows current standards in major university hospitals performing this technique. Furthermore, preliminary data also suggest efficacy and safety for patients treated with SBRT for spinal metastases in a previously radiated field. However, well defined prospective outcomes are lacking in this patient group.

There a 3 cohorts for this study each with a target accrual of 30 patients. Cohort 1: patients with spinal metastases and no prior radiation.

Cohort 2: patients with spinal metastases with a history of previous radiation to the affected spinal segment.

Cohort 3: post-operative patients with spinal metastases with or without a history of previous radiation to the affected spinal segment.

All patients will be treated with either 20-24 Gy in one fraction (recommended) or 20-24 Gy in two fractions, or 20-24 Gy in three fractions. There is also and optional imaging component of this study.

The purpose of the study is to determine the efficacy of spine SBRT in select groups of patients using image based and symptom based local control criteria

ELIGIBILITY:
Inclusion Criteria:

* Solitary or oligometastatic spine disease (maximum 5 sites of metastases), or bone only metastatic disease (regardless of the number) in otherwise high performance status patients, or patients with diffuse metastatic disease where the patient survival is expected to be at least 6 months
* Maximum of 2 consecutive spinal segments involved by tumor for treatment otherwise a maximum of 3 sites within the spine to be treated in a single session
* Previously irradiated: up to one course where the maximum BED previously delivered is no more than 100 Gy2 (50 Gy2/2) and >5 month interval from prior radiation to planned SBRT (Cohort 2) or first part of cohort 3
* Karnofsky Performance Status >60
* Had an MRI or CT documented spinal tumor and MRI of full spine no more than 8 weeks prior to SBRT (if patients cannot have a MRI then a CT myelogram is required)
* Had a histological confirmation of neoplastic disease
* Expected to have survival of > 3 months regardless of the number of metastases
* Able to lie still and in a supine position on the treatment couch for up to 1 hour
* Age >18
* Adequate Bowel or urinary function

Exclusion Criteria:

* A Pacemaker such that MRI cannot be performed or the treatment cannot be delivered safely
* Scleroderma or connective tissue disease as a contra-indication to radiotherapy
* Unable to lie supine (i.e. tolerate treatment)
* Previously treated with any radionuclides within 30 days prior to SBRT
* Had external beam radiotherapy to the same area less than 5 months prior to SBRT and/or a course of radiation previously delivered >100 Gy2 (50 Gy2/2)
* Significant or progressive neurologic deficit
* Malignant epidural spinal cord compression or cauda equina syndrome
* Spine instability, or neurological deficit resulting from bony compression of neural structures
* Receiving chemotherapy for at least 1 week prior to SBRT and chemotherapy for one week following SBRT
* Expected patient survival < 3 months

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2011-06; Primary Completion 2015-12 (Actual); Study Completion 2017-04-27 (Actual)

PRIMARY OUTCOMES:
To determine the efficacy of spine SBRT in select groups of patients using image based and symptom based local control criteria | 5 years

SECONDARY OUTCOMES:
To determine prospective pain and functional outcome data using the Brief Pain Inventory questionnaire | 5 years
To prospectively document quality of life outcomes for patients post-SBRT using the validated EORTC QLQ - BM22 and C-15 PAL | 5 years
To determine pain flare prospective data by using the Pain Diary for first 10 days after radiation. | 5 years
To prospectively evaluate neurologic outcomes using the ASIA questionnaire | 5 years
To evaluate acute and late toxicity of RT using NCIC Common Toxicity Criteria v. 3.0 | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: John Cho, MD, Principal Investigator — University Health Network, Princess Margaret Hospital
Locations (1):
- University Health Network, Princess Margaret Hospital, Toronto, Ontario, Canada